CLINICAL TRIAL: NCT00620867
Title: A Study of the Efficacy and Tolerability of Once Daily Celebrex (Celecoxib) and Three Times Daily Ibuprofen vs. Placebo in the Treatment of Subjects With Osteoarthritis of the Knee
Brief Title: Efficacy and Safety of Celecoxib Versus Ibuprofen in the Treatment of Osteoarthritis of the Knee (United States)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3191063
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ibuprofen; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ibuprofen (Experimental)
  Interventions: Drug: Ibuprofen
- Celecoxib (Experimental)
  Interventions: Drug: celecoxib
- placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Ibuprofen — 800 mg oral tablet three time daily with meals for 6 weeks
  Arms: Ibuprofen
Drug: celecoxib — 200 mg oral capsule once daily with morning meal for 6 weeks
  Arms: Celecoxib
Other: placebo — matched placebo orally for 6 weeks
  Arms: placebo

SUMMARY:
To compare the efficacy and safety of celecoxib versus ibuprofen in subjects with osteoarthritis (OA) of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Aged >= 40 years old
* Diagnosed with OA of the knee according to the American College of Rheumatology and OA in flare state at baseline visit
* Functional capacity class of I-III

Exclusion Criteria:

* Inflammatory arthritis or gout or pseudo-gout with acute flare within the past 2 years (subjects with fibrositis or fibromyalgia will not be excluded)
* Acute joint trauma at index joint within the past 3 months with active symptoms
* Score of >=20 on PHQ-9 or score of >=1 on PHQ-9 item i
* Use of mobility assisting device for <6 weeks or use of walker

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2002-10; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in patient's assessment of arthritis pain according to visual analogue scale (VAS) | Week 6

SECONDARY OUTCOMES:
Vital signs | Weeks 2 and 6
Physical examination | Week 6
Laboratory test results | Week 6
Adverse events | Weeks 2 and 6
Change from baseline in patient's and physician's global assessment of pain | Weeks 2 and 6
Pain Satisfaction Scale | Days 1-7
Change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index | Week 6
Patient Health Questionnaire (PHQ-9) | Week 6
Change from baseline in patient's assessment of arthritis pain according to VAS | Week 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- United States (33):
  - Pfizer Investigational Site, Anniston, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Paramount, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Edison, New Jersey
  - Pfizer Investigational Site, South Plainfield, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Jenkintown, Pennsylvania
  - Pfizer Investigational Site, Newtown, Pennsylvania
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Johnson City, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Layton, Utah
  - Pfizer Investigational Site, Danville, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191063&StudyName=Efficacy%20and%20Safety%20of%20Celecoxib%20versus%20Ibuprofen%20in%20the%20Treatment%20of%20Osteoarthritis%20of%20the%20Knee%20%28United%20States%29